CLINICAL TRIAL: NCT05939518
Title: The Contribution of Liberal Fluid Therapy to Glycocalyx Shedding, Interstitial Edema and Fluid Accumulation During Moderate Surgery
Brief Title: Fluid Therapy and Glycocalyx Shedding During Moderate Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 0388-19-HMO; 008932_2020-05-12_MOH (Registry Identifier: Israeli Ministry of Health)
Record Dates: First submitted 2023-06-15; First posted 2023-07-11 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Abdominoplasty
Keywords: Glycocalyx; IV Fluids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liberal Lactated Ringer Fluid Protocol with Ephedrine and Phenylephrine Boluses (Experimental): IV Infusion of 500 ml of lactated Ringer's (RL) solution during the induction of anesthesia followed by an infusion of RL at a rate of 8.0 ml/kg/h throughout the maintenance phase of anesthesia. The anesthesia care provider will be allowed free use of IV boluses of ephedrine or phenylephrine to target a mean arterial blood pressure of >60 mmHg.
  Interventions: Other: Lactated Ringer's Fluid Bolus Response to Low Urinary Output; Other: Post-Anesthesia Care Unit Lactated Ringer's Fluid Management Protocol
- Restrictive Lactated Ringer Fluid Protocol with Noradrenaline Infusion (Active Comparator): IV Infusion of 200 ml of lactated Ringer's (RL) solution during the induction of anesthesia followed by an infusion of RL at a rate of 2.0 ml/kg/h + an infusion of noradrenaline throughout the maintenance phase of anesthesia, through a large peripheral vein. The noradrenaline infusion rate will be titrated after an initial bolus of 10 μg, from an initial rate of 2.0 μg/kg/h, which may be raised up to 8.0 μg/kg/h, to target a mean arterial blood pressure (MBP) of >60 mmHg. If the MBP target is still not achieved, the RL infusion rate may be increased up to 4.0 ml/kg/h.
  Interventions: Other: Lactated Ringer's Fluid Bolus Response to Low Urinary Output; Other: Post-Anesthesia Care Unit Lactated Ringer's Fluid Management Protocol

INTERVENTIONS:
Other: Lactated Ringer's Fluid Bolus Response to Low Urinary Output — During the surgical procedure and the subsequent stay in the Post-Anesthesia Care Unit: if the study participant's urine output (UO) remains <0.3 ml/kg/h for two consecutive hours, an IV bolus of 250 ml of lactated Ringer's solution will be administered over 15 min and repeated every 30 min until the UO reaches >0.3 ml/kg/h.
Other: Post-Anesthesia Care Unit Lactated Ringer's Fluid Management Protocol — During their stay in the Post-Anesthesia Care Unit, patients will receive a 1.5 ml/kg/h IV infusion of lactated Ringer's solution.
  Other Names: Recovery Room Fluid Management Protocol

SUMMARY:
Goal-directed fluid therapy is one of the most accepted strategies in intraoperative fluid therapy, although potential fluid overload is a possible drawback. Fluid overload has recently been shown to cause damage to the glycocalyx and to increase extravasation of fluids into the interstitial space.

This study aims to determine whether liberal fluid administration during moderate surgery results in impairment to the endothelial glycocalyx and causes edema.

Participants will be randomized to receive either a liberal or restrictive fluid protocol with vasopressor support. The investigators will measure interstitial edema by clinical signs, pulmonary congestion by ultrasound, and extracellular water by bioimpedance. Impairment of glycocalyx will be estimated by measuring blood levels of shedding markers. In addition, wound healing and early postoperative outcome will be estimated by POMS.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for abdominoplasty.
* American Society of Anesthesiologists Classification 1 or 2.

Exclusion Criteria:

* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change from preoperative serum concentration of Heparan Sulfate. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Change from preoperative serum concentration of Syndecan-1. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Change from preoperative serum concentration of Hyaluronic Acid. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Change from preoperative serum concentration of Sphingosine-1-Phosphate. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Appearance of B-lines on lung ultrasonography. | Two hours after completion of surgery.
  Bilateral ultrasonography of the study participant's lungs, performed by a physician using two views: posterior and lateral.
Early appearance of peripheral pitting edema. | Two hours after completion of surgery.
  Bilateral physical examination of the study participant's wrists and ankles, performed by a physician.
Late appearance of peripheral pitting edema. | During the first postoperative day.
  Bilateral physical examination of the study participant's wrists and ankles, performed by a physician.
Postoperative Morbidity Survey (POMS) Score. | During the first postoperative day.
  Clinically evaluated by a physician for each study participant.
Early change in the percentage of Total Body Water and Extracellular Water. | Immediately after completion of surgery.
  Measured by bioimpedance using a commercially available device connected to the study participant.
Late change in the percentage of Total Body Water and Extracellular Water. | Two hours after completion of surgery.
  Measured by bioimpedance using a commercially available device connected to the study participant.

SECONDARY OUTCOMES:
Change from preoperative body weight. | During the first postoperative day.
  Recorded while the study participant stands on an electronic scale.
Volume of urine produced during the procedure. | Immediately after completion of surgery.
  Measured using a volumetric graduated urine collection container connected to a Foley catheter placed in the urinary bladder of the study participant.
Change from preoperative Heart Rate. | Immediately after completion of surgery.
  Measured using a continuous electrocardiography monitor connected to the study participant.
Change from preoperative Mean Arterial Blood Pressure. | Immediately after completion of surgery.
  Measured using an automated oscillometric blood pressure monitoring device with its cuff placed on one of the arms of the study participant.
Early change from preoperative Cardiac Output. | Immediately after completion of surgery.
  Measured non-invasively using a commercially available device connected to the study participant.
Late change from preoperative Cardiac Output. | Two hours after completion of surgery.
  Measured non-invasively using a commercially available device connected to the study participant.
Early change from preoperative serum concentration of C-Reactive Protein. | Immediately after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Late change from preoperative serum concentration of C-Reactive Protein. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Early change from preoperative serum concentration of Lactate. | Immediately after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Late change from preoperative serum concentration of Lactate. | Two hours after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Change from preoperative serum concentration of Creatinine. | Immediately after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.
Change from preoperative serum concentration of Hemoglobin. | Immediately after completion of surgery.
  Measured using blood samples drawn from a peripheral vein of the study participant and analyzed in a laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Galel Yakobi, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Ein-Carem Medical Center, Jerusalem, Israel